CLINICAL TRIAL: NCT03755999
Title: A Cue-based Developmental Approach Toward the Preterm Infants During Feeding Transition Period - Explore Clinical Facts, Evaluate Intervention Effects and Develop Clinical Guideline
Brief Title: A Cue-based Developmental Approach Toward the Preterm Infants During Feeding Transition Period
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MOST 107-2314-B-006-009-MY3
Record Dates: First submitted 2018-08-22; First posted 2018-11-28 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-07

CONDITIONS: Preterm Infant; Feeding Behavior; Feeding Patterns
Keywords: preterm infants; transitional feeding period; cue-based care; clinical guidelines
MeSH Terms: conditions — Premature Birth; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIOMI treat group (Experimental): Preterm infant receive oral massage using the premature infant oral motor intervention (PIOMI)
  Interventions: Other: The premature infant oral motor intervention (PIOMI)
- Routine care group (No Intervention): Preterm infant receive routine care of neonatal intensive care unit(NICU)

INTERVENTIONS:
Other: The premature infant oral motor intervention (PIOMI) — The premature infant oral motor intervention (PIOMI) is an oral motor program that provides assisted movement to activate muscle contraction and provides movement against resistance to build strength in the areas of the mouth necessary for feeding. It is designed to increase the maturation of neural structures, improving their ability to suck and swallow.
  Other Names: Cue-based feeding
  Arms: PIOMI treat group

SUMMARY:
The coordination of sucking, swallowing, and breathing during the transition from gavage to oral feeding is a challenge for preterm infants. Efficient management of the feeding transition without other comorbidities can not only improve their oral movements and gastrointestinal function development, facilitate their oral feeding learning behavior, but also facilitate them to direct breastfeeding, improve mother-infant attachment, and ultimately reduce the length of hospitalization. However, the current status of strategies in supporting preterm infants throughout their feeding transition are inconsistent, and lack of guidelines and monitor indicators based on existing evidence.

This project proposed a three-year plan the explore the current situation, examine effective strategies for care bundles, and further develop a new clinical guideline that can be implemented in the future. The first year of this research will use chart review among two neonatal intensive care units of Medical Center from Taipei and Tainan. A semi-structured interview and questionnaire (DSCS-N) will be used to explore nurses' knowledge, attitude and skills of developmental care; and the experience of caring for preterm infants during feeding transition in the neonatal intensive care units. In addition, gestational age, body weight, gavage and oral feeding amount, and special events happened during feeding will be recorded and analyzed.

The second year, an experimental with a stratified random assignment and repeated measure design will be used with feeding transition care bundles. 120 preterm infants will be recruited and assigned to experimental or control group. The subjects will be fed by the routine care approach or by the feeding transition approach in one neonatal intensive care unit. Intervention components include oral stimulation and cue-based feeding during the transition to oral feeding. Study measures will include physical indicators, POFRAS and EFS during feeding to evaluate the implementation and guide further development of the clinical guideline.

The third year of guideline development will follow Bowker and the National Health Insurance Bureau which including 5 stage. The results of this guideline can offer better recommendations to support preterm infants' oral development, provide cue-based feeding, and help them succeed in the transition to oral nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infant born less then 33 weeks
* Fraction of inspired oxygen(FiO2) less then 30%
* Can tolerance enteral feeding

Exclusion Criteria:

* Using ventilator(except non-invasive ventilator)
* Complications including Hypoxic Ischemic Encephalopathy (HIE), Intraventricular Hemorrhage (IVH) ≥Grade III, Periventricular Leukomalacia (PVL), Necrotizing Enterocolitis(NEC) ≥Stage II
* Congenital abnormalities including chromosomal abnormalities, congenital anomalies of digestive system, cleft lip and palate
* Because of custody problem or can't get the inform consent of the preterm infant's parents/guardian

Max Age: 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Preterm infant's oral feeding readiness | Change from day 1(Baseline) up to day 7 in oral stimulation phase
  We use the Preterm Oral Feeding Readiness Assessment Scales (POFRAS) to assess preterm infants' readiness to start oral feeding. The scale comprised of 5 five categories including corrected Gestational Age, Behavioral Organization (3 item), Oral Posture (2 item), Oral Reflexes (4 item), Nonnutritive Sucking (8 item) with a total of 18 items to evaluate. Each item score from 0~2, the higher the score means that the preterm infant has better oral feeding preparation.
Preterm infant's oral feeding skills | From day 1(Baseline) up to the day 30 in cue-base feeding phase
  Using Early Feeding Skills Assessments for Preterm Infants (EFS). The Early Feeding Skills Assessments for Preterm Infants (EFS) checklist is to assess preterm infants' oral feeding readiness (before feeding; yes/no), oral feeding skill (when feeding; all/most/some/none; never/occasionally/often), oral feeding tolerance (after feeding; yes/no) and feeding descriptors(after feeding).

SECONDARY OUTCOMES:
Body weight change | Change from day 1(baseline) up to the day 200.
  body weight change in grams
hospital stay length(days) | From day 1 up to the day 200.
  How many days from admission(birth day) to discharge(leave) hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Chih Huang, Principal Investigator — Department of Nursing, College of Medicine, National Cheng-Kung University
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

REFERENCES:
- [Background] Aita M, Snider L. The art of developmental care in the NICU: a concept analysis. J Adv Nurs. 2003 Feb;41(3):223-32. doi: 10.1046/j.1365-2648.2003.02526.x. PMID 12581110
- [Background] Als H. Toward a synactive theory of development: Promise for the assessment and support of infant individuality. Infant Mental Health Journal 3(4): 229-243, 1982.
- [Background] Als H, Butler S, Kosta S, McAnulty G. The Assessment of Preterm Infants' Behavior (APIB): furthering the understanding and measurement of neurodevelopmental competence in preterm and full-term infants. Ment Retard Dev Disabil Res Rev. 2005;11(1):94-102. doi: 10.1002/mrdd.20053. PMID 15856436
- [Background] Bala P, Kaur R, Mukhopadhyay K, Kaur S. Oromotor Stimulation for Transition from Gavage to Full Oral Feeding in Preterm Neonates: A Randomized controlled trial. Indian Pediatr. 2016 Jan;53(1):36-8. doi: 10.1007/s13312-016-0786-3. PMID 26840669
- [Background] Balshem H, Helfand M, Schunemann HJ, Oxman AD, Kunz R, Brozek J, Vist GE, Falck-Ytter Y, Meerpohl J, Norris S, Guyatt GH. GRADE guidelines: 3. Rating the quality of evidence. J Clin Epidemiol. 2011 Apr;64(4):401-6. doi: 10.1016/j.jclinepi.2010.07.015. Epub 2011 Jan 5. PMID 21208779
- [Background] Bolzan Gde P, Berwig LC, Prade LS, Cuti LK, Yamamoto RC, Silva AM, Weinmann AR. Assessment for oral feeding in preterm infants. Codas. 2016 Jul 4;0:0. doi: 10.1590/2317-1782/20162015115. English, Portuguese. PMID 27383226
- [Background] Brouwers MC, Kho ME, Browman GP, Burgers JS, Cluzeau F, Feder G, Fervers B, Graham ID, Grimshaw J, Hanna SE, Littlejohns P, Makarski J, Zitzelsberger L; AGREE Next Steps Consortium. AGREE II: advancing guideline development, reporting and evaluation in health care. CMAJ. 2010 Dec 14;182(18):E839-42. doi: 10.1503/cmaj.090449. Epub 2010 Jul 5. No abstract available. PMID 20603348
- [Background] Byers JF. Components of developmental care and the evidence for their use in the NICU. MCN Am J Matern Child Nurs. 2003 May-Jun;28(3):174-80; quiz 181-2. doi: 10.1097/00005721-200305000-00007. PMID 12771696
- [Background] Fujinaga CI, Zamberlan NE, Rodarte MD, Scochi CG. [Reliability of an instrument to assess the readiness of preterm infants for oral feeding]. Pro Fono. 2007 Apr-Jun;19(2):143-50. doi: 10.1590/s0104-56872007000200002. Portuguese. PMID 17710340
- [Background] da Costa SP, van der Schans CP. The reliability of the Neonatal Oral-Motor Assessment Scale. Acta Paediatr. 2008 Jan;97(1):21-6. doi: 10.1111/j.1651-2227.2007.00577.x. PMID 18201309
- [Background] da Costa SP, Hubl N, Kaufman N, Bos AF. New scoring system improves inter-rater reliability of the Neonatal Oral-Motor Assessment Scale. Acta Paediatr. 2016 Aug;105(8):e339-44. doi: 10.1111/apa.13461. Epub 2016 Jun 6. PMID 27164051
- [Background] Fucile S, Gisel EG, Lau C. Effect of an oral stimulation program on sucking skill maturation of preterm infants. Dev Med Child Neurol. 2005 Mar;47(3):158-62. doi: 10.1017/s0012162205000290. PMID 15739719
- [Background] Fucile S, Gisel E, Lau C. Oral stimulation accelerates the transition from tube to oral feeding in preterm infants. J Pediatr. 2002 Aug;141(2):230-6. doi: 10.1067/mpd.2002.125731. PMID 12183719
- [Background] Fujinaga CI, de Moraes SA, Zamberlan-Amorim NE, Castral TC, de Almeida e Silva A, Scochi CG. Clinical validation of the Preterm Oral Feeding Readiness Assessment Scale. Rev Lat Am Enfermagem. 2013 Jan-Feb;21 Spec No:140-5. doi: 10.1590/s0104-11692013000700018. English, Portuguese. PMID 23459901
- [Background] Gennattasio A, Perri EA, Baranek D, Rohan A. Oral feeding readiness assessment in premature infants. MCN Am J Matern Child Nurs. 2015 Mar-Apr;40(2):96-104; E9-10. doi: 10.1097/NMC.0000000000000115. PMID 25494013
- [Background] Greene Z, O'Donnell CP, Walshe M. Oral stimulation for promoting oral feeding in preterm infants. Cochrane Database Syst Rev. 2016 Sep 20;9(9):CD009720. doi: 10.1002/14651858.CD009720.pub2. PMID 27644167
- [Background] Griffith T, Rankin K, White-Traut R. The Relationship Between Behavioral States and Oral Feeding Efficiency in Preterm Infants. Adv Neonatal Care. 2017 Feb;17(1):E12-E19. doi: 10.1097/ANC.0000000000000318. PMID 27649302
- [Background] Jones LR. Oral feeding readiness in the neonatal intensive care unit. Neonatal Netw. 2012 May-Jun;31(3):148-55. doi: 10.1891/0730-0832.31.3.148. PMID 22564310
- [Background] Kirk AT, Alder SC, King JD. Cue-based oral feeding clinical pathway results in earlier attainment of full oral feeding in premature infants. J Perinatol. 2007 Sep;27(9):572-8. doi: 10.1038/sj.jp.7211791. Epub 2007 Jul 12. PMID 17625573
- [Background] Kish MZ. Oral feeding readiness in preterm infants: a concept analysis. Adv Neonatal Care. 2013 Aug;13(4):230-7. doi: 10.1097/ANC.0b013e318281e04e. PMID 23912014
- [Background] Kim JS, Shin HS. [Development of the Developmental Support Competency Scale for Nurses Caring for Preterm Infants]. J Korean Acad Nurs. 2016 Dec;46(6):793-803. doi: 10.4040/jkan.2016.46.6.793. Korean. PMID 28077827
- [Background] Lapillonne A. Enteral and parenteral lipid requirements of preterm infants. World Rev Nutr Diet. 2014;110:82-98. doi: 10.1159/000358460. Epub 2014 Apr 11. PMID 24751623
- [Background] Lau C. Development of infant oral feeding skills: what do we know? Am J Clin Nutr. 2016 Feb;103(2):616S-21S. doi: 10.3945/ajcn.115.109603. Epub 2016 Jan 20. PMID 26791183
- [Background] Lau C, Smith EO, Schanler RJ. Coordination of suck-swallow and swallow respiration in preterm infants. Acta Paediatr. 2003 Jun;92(6):721-7. PMID 12856985
- [Background] Leite HP. Adequate nutrition can improve the outcome of premature infants. Rev Bras Ter Intensiva. 2011 Dec;23(4):391-3. No abstract available. English, Portuguese. PMID 23949452
- [Background] Liaw JJ, Chen SY, Yin YT. Nurses' beliefs and values about doing cue-based care in an NICU in Taiwan. J Nurs Res. 2004 Dec;12(4):275-86. doi: 10.1097/01.jnr.0000387512.36996.4c. PMID 15619178
- [Background] Lima AH, Cortes MG, Bouzada MC, Friche AA. Preterm newborn readiness for oral feeding: systematic review and meta-analysis. Codas. 2015 Jan-Feb;27(1):101-7. doi: 10.1590/2317-1782/20152014104. English, Portuguese. PMID 25885204
- [Background] Lubbe W. Clinicians guide for cue-based transition to oral feeding in preterm infants: An easy-to-use clinical guide. J Eval Clin Pract. 2018 Feb;24(1):80-88. doi: 10.1111/jep.12721. Epub 2017 Mar 2. PMID 28251754
- [Background] McCain GC. An evidence-based guideline for introducing oral feeding to healthy preterm infants. Neonatal Netw. 2003 Sep-Oct;22(5):45-50. doi: 10.1891/0730-0832.22.5.45. PMID 14598979
- [Background] McClure RJ. Trophic feeding of the preterm infant. Acta Paediatr Suppl. 2001 Mar;90(436):19-21. doi: 10.1111/j.1651-2227.2001.tb01623.x. PMID 11332950
- [Background] McInnes RJ, Shepherd AJ, Cheyne H, Niven C. Infant feeding in the neonatal unit. Matern Child Nutr. 2010 Oct;6(4):306-17. doi: 10.1111/j.1740-8709.2009.00210.x. PMID 21050385
- [Background] Newland L, L'huillier MW, Petrey B. Implementation of cue-based feeding in a level III NICU. Neonatal Netw. 2013 Mar-Apr;32(2):132-7. doi: 10.1891/0730-0832.32.2.132. No abstract available. PMID 23477983
- [Background] Otto DM, de Almeida ST. Oral feeding performance in premature infants stimulated by swallowing technical training. Audiology - Communication Research 22: e1717, 2017.
- [Background] Pados BF, Park J, Estrem H, Awotwi A. Assessment Tools for Evaluation of Oral Feeding in Infants Younger Than 6 Months. Adv Neonatal Care. 2016 Apr;16(2):143-50. doi: 10.1097/ANC.0000000000000255. PMID 26945280
- [Background] Pickler RH, Wetzel PA, Meinzen-Derr J, Tubbs-Cooley HL, Moore M. Patterned feeding experience for preterm infants: study protocol for a randomized controlled trial. Trials. 2015 Jun 4;16:255. doi: 10.1186/s13063-015-0781-3. PMID 26041365
- [Background] Porges SW. The polyvagal perspective. Biol Psychol. 2007 Feb;74(2):116-43. doi: 10.1016/j.biopsycho.2006.06.009. Epub 2006 Oct 16. PMID 17049418
- [Background] Ross ES, Philbin MK. Supporting oral feeding in fragile infants: an evidence-based method for quality bottle-feedings of preterm, ill, and fragile infants. J Perinat Neonatal Nurs. 2011 Oct-Dec;25(4):349-57; quiz 358-9. doi: 10.1097/JPN.0b013e318234ac7a. PMID 22071619
- [Background] Shaker CS. Cue-based feeding in the NICU: using the infant's communication as a guide. Neonatal Netw. 2013 Nov-Dec;32(6):404-8. doi: 10.1891/0730-0832.32.6.404. PMID 24195800
- [Background] Simpson C, Schanler RJ, Lau C. Early introduction of oral feeding in preterm infants. Pediatrics. 2002 Sep;110(3):517-22. doi: 10.1542/peds.110.3.517. PMID 12205253
- [Background] Swant L, Fairchild R. Placing the bottle or breast in their premature hands: A review of cue-based feeding research. Journal of Neonatal Nursing 20(3): 122-128, 2014.
- [Background] Thomas JA. Guidelines for bottle feeding your premature baby. Adv Neonatal Care. 2007 Dec;7(6):311-8. doi: 10.1097/01.ANC.0000304971.69578.f7. PMID 18097214
- [Background] Thoyre SM, Shaker CS, Pridham KF. The early feeding skills assessment for preterm infants. Neonatal Netw. 2005 May-Jun;24(3):7-16. doi: 10.1891/0730-0832.24.3.7. PMID 15960007
- [Background] Tian X, Yi LJ, Zhang L, Zhou JG, Ma L, Ou YX, Shuai T, Zeng Z, Song GM. Oral Motor Intervention Improved the Oral Feeding in Preterm Infants: Evidence Based on a Meta-Analysis With Trial Sequential Analysis. Medicine (Baltimore). 2015 Aug;94(31):e1310. doi: 10.1097/MD.0000000000001310. PMID 26252313
- [Background] Touzet S, Beissel A, Denis A, Pillet F, Gauthier-Moulinier H, Hommey S, Claris O; TOP Study Group. Effectiveness of a nurse educational oral feeding programme on feeding outcomes in neonates: protocol for an interrupted time series design. BMJ Open. 2016 Apr 15;6(4):e010699. doi: 10.1136/bmjopen-2015-010699. PMID 27084282
- [Background] White A, Parnell K. The transition from tube to full oral feeding (breast or bottle) - A cue-based developmental approach. Journal of Neonatal Nursing 19(4): 189-197, 2013.
- [Background] Younesian S, Yadegari F, Soleimani F. Impact of Oral Sensory Motor Stimulation on Feeding Performance, Length of Hospital Stay, and Weight Gain of Preterm Infants in NICU. Iran Red Crescent Med J. 2015 Jul 31;17(7):e13515. doi: 10.5812/ircmj.17(5)2015.13515. eCollection 2015 Jul. PMID 26421163
- [Background] Ziadi M, Héon M, Aita M. A critical review of interventions supporting transition from gavage to direct breastfeeding in hospitalized preterm infants. Newborn and Infant Nursing Reviews 16(2): 78-91, 2016.
- [Background] Lin CH, Chang YJ, Lin CN, Huang MC. [Feeding preterm infants: application of developmental care]. Hu Li Za Zhi. 2012 Jun;59(3):107-12. Chinese. PMID 22661039
- [Background] Lin SC, Lin CH, Zhang JW, Chen SM, Chen CL, Huang MC. [Breast- and bottle-feeding in preterm infants: a comparison of behavioral cues]. Hu Li Za Zhi. 2013 Dec;60(6):27-34. doi: 10.6224/JN.60.6.27. Chinese. PMID 24310551
- [Background] Chang YW, Chang YJ. [The relationship between oral feeding and cardiorespiratory regulation of premature infants]. Hu Li Za Zhi. 2008 Jun;55(3):5-10. Chinese. PMID 18543179